CLINICAL TRIAL: NCT03434574
Title: Evaluation of the Effect of Chokeberry (Aronia Melanocarpa) Polyphenols on Blood Pressure in Prehypertensive Healthy Men and Women
Brief Title: Aronia Berry Consumption on Blood Pressure
Acronym: ABP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Naturex-Dbs (Industry)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Principal investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Aronia BP
Record Dates: First submitted 2018-01-11; First posted 2018-02-15 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Prehypertension; Healthy
Keywords: (Poly)phenols; Aronia berry; Blood pressure; Vascular function
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Formulation containing inert artificially colored maltodextrin, once daily, in a 1-hard capsule regimen (500 mg)
  Interventions: Dietary Supplement: Placebo
- Aronia extract (Active Comparator): Formulation of an aronia extract ingredient in a 1-hard capsule regimen (500 mg)
  Interventions: Dietary Supplement: Aronia extract

INTERVENTIONS:
Dietary Supplement: Placebo — Identical formulation as the treatment consisting of colored maltodextrin using artificial colors.
  Arms: Placebo
Dietary Supplement: Aronia extract — Powdered extract obtained from aronia berries (Aronia melanocarpa).
  Arms: Aronia extract

SUMMARY:
Aronia berries are a native North American berry with high naturally occurring anthocyanins among other polyphenols. Based on their polyphenol composition, there is growing interest in the potential for Aronia berries to elicit health promoting cardio-metabolic effects. Specifically, Aronia berry extracts, which provide a concentrated source of polyphenols, may improve blood vessel function.

Thus, the primary focus of this project is to evaluate the effects of Aronia berry polyphenols on blood pressure and other biomarkers of cardiovascular disease risk such as endothelial function, arterial stiffness and blood lipids.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 40-70 years old
* Blood pressure comprised between: SBP 120/139 mmHg or DBP 80/89 mmHg
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
* Are able to understand the nature of the study
* Able and willing to give signed written informed consent
* Signed informed consent form

Exclusion Criteria:

* Manifest cardiovascular disease including coronary artery disease, cerebrovascular disease and peripheral artery disease
* Grade 1 hypertensive or above, as defined as SBP superior or equal to 140 mmHg or DBP superior or equal to 90 mmHg
* Obese participants, defined as BMI superior or equal to 30
* Diabetes mellitus and metabolic syndrome
* Acute inflammation
* Chronic and acute disease
* Terminal renal failure and other kidney abnormalities
* Malignancies
* Abnormal heart rhythm
* Allergies to berries or other significant food allergy.
* Subjects who require treatment for hypertension at any time (e.g. statins, aspirin, blood pressure lowering drugs)
* Subjects who took food supplements, dietary supplement or herbal remedies within 1 month of study start
* Subjects who have lost more than 10% of their weight in the past 6 months or are currently in a diet
* Subjects who reported participant in another study within 1 month before the study start
* Subjects who smoke an irregular amount of cigarettes per day
* Subjects who require chronic antimicrobial or antiviral treatment
* Subjects with unstable psychological condition
* Subjects with history of cancer, myocardial infarction, cerebrovascular incident
* Unable to swallow the capsule
* Pregnant, lactating or planning to become pregnant, as well as premenopausal women who do not have an adequate method of contraception
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline ambulatory blood pressure after 12-week consumption | Baseline and 12 weeks
  Determine the effect of the Aronia extract vs Placebo on ambulatory 24-hour systolic and diastolic blood pressure at 12 weeks post consumption, compared to the baseline.

SECONDARY OUTCOMES:
Office blood pressure | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Determine the effect of the Aronia extract vs Placebo on office systolic and diastolic blood pressure, at 12 weeks post consumption
Heart rate | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Determine the effect of the Aronia extract vs Placebo on heart rate, at 12 weeks post consumption
Flow-mediated dilation | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Determine the effect of the Aronia extract vs Placebo on flow-mediated dilation at 12 weeks post consumption
Blood flow velocity | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Determine the effect of the Aronia extract vs Placebo on blood flow velocity at 12 weeks post consumption
Pulse wave velocity (PWV) | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Determine the effect of the Aronia extract vs Placebo on pulse wave velocity (PWV) using a Sphygmocor device, at 12 weeks post consumption
Augmentation Index (AIx) | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Determine the effect of the Aronia extract vs Placebo on augmentation Index (AIx) using a Sphygmocor device, at 12 weeks post consumption
Blood lipids | Baseline and 12 weeks
  Determine the effect of the Aronia extract vs Placebo on blood lipids (Total, HDL and LDL cholesterol, triglycerides), at 12 weeks post consumption
Blood cortisol | Baseline and 12 weeks
  Determine the effect of the Aronia extract vs Placebo on blood cortisol levels, at 12 weeks post consumption
Number of volunteers with treatment-related adverse events | Baseline and 12 weeks
  The number of volunteers with treatment-related adverse events will be assessed by questionnaires and interviews.
24-hour heart rate | Baseline and 12 weeks
  Determine the effect of the Aronia extract vs Placebo on 24-hour heart rate, using a monitor, at 12 weeks post consumption

OTHER OUTCOMES:
Plasma aronia berry (poly)phenol metabolites | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Measured by liquid chromotography- mass spectrometry (LC/MS) 0 and 2 hours postconsumption at day 1 (baseline) and after 12 weeks.
Microbiome analysis | Baseline and 12 weeks
  Stool sample collection (Omnigene gut collection kit)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Department of Life Sciences and Medecine, London, Central London
  - King's College London, London, England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Sayec M, Xu Y, Laiola M, Gallego FA, Katsikioti D, Durbidge C, Kivisild U, Armes S, Lecomte M, Fanca-Berthon P, Fromentin E, Plaza Onate F, Cruickshank JK, Rodriguez-Mateos A. The effects of Aronia berry (poly)phenol supplementation on arterial function and the gut microbiome in middle aged men and women: Results from a randomized controlled trial. Clin Nutr. 2022 Nov;41(11):2549-2561. doi: 10.1016/j.clnu.2022.08.024. Epub 2022 Sep 6. PMID 36228567